CLINICAL TRIAL: NCT03837834
Title: Effects of 6 Weeks High-intensity Interval Training on Muscle Strength and Cardiorespiratory Response Among Spinal Cord Injury
Brief Title: Effects of 6 Weeks High-intensity Interval Training Among Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, MOHD KHAIRUL AZHAR BIN ARIFFIN, Principal Investigator, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201682-4100
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: INCOMPLETE SPINAL CORD INJURY (ASIA D)
Keywords: HIGH INTENSITY INTERVAL TRAINING; INCOMPLETE SPINAL CORD INJURY; MUSCLE STRENGTH; CARDIO-RESPIRATORY FITNESS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 MIN X 4 MIN HIIT of FES-LCE (Experimental): 4 min of high-intensity phase intersperses with 4 min of low-intensity phase for a total of 5 bouts.
  Interventions: Other: Functional Electrical Stimulation Leg Cycling Exercise
- 2 MIN X 2 MIN HIIT of FES-LCE (Experimental): 2 min of high-intensity phase intersperses with 2 min of low-intensity phase for a total of 10 bouts.
  Interventions: Other: Functional Electrical Stimulation Leg Cycling Exercise

INTERVENTIONS:
Other: Functional Electrical Stimulation Leg Cycling Exercise — FES- leg cycling for 45 minutes (3 min warm up + 40 min HIIT + 2 min cooldown). The FES will be applied via surface electrodes and the stimulation intensity based on your tolerance level.

SUMMARY:
The training consists of 6 weeks of functional electrical stimulation leg cycling exercise (FES-LCE) program. The training program comprises of 2 visits per week. Each visit consists of FES-LCE for 45 minutes. Throughout the 6 weeks program, there will be testing/assessment sessions on week 1, week 3 and week 6. The FES will be applied via surface electrodes and the stimulation intensity based on the participant's tolerance level.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with incomplete spinal cord injury (SCI) at least one year prior to participation.
* Age between 18-75 years old.
* Both male and female.
* Have at least 90º bilateral knee flexion.
* Moderate neurological induce weakness in quadriceps muscle of 1 leg that is responsive to electrical stimulation (moderate weakness was defined as 3/5 or 4/5 on manual muscle testing).
* Able to perform cycling activity.
* Normal upper limb function.
* Able to follow command.

Exclusion Criteria:

* Had a recent history of trauma to the lower limb.
* Severely infected skin pressure sore on weight-bearing skin areas.
* Illness caused by acute urinary tract infection.
* Uncontrolled spasticity or pain.
* History of cardiovascular/cardiorespiratory problem.
* Orthostatic hypotension.
* Unhealed decubiti at electrode placement area.
* Recurrent autonomic dysreflexia.
* Active heterotopic ossification.
* Other peripheral or central neurologic injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Changes of peak torque of Quadriceps and Hamstring | Changes of peak torque at 6 week
  Isometric peak torque for quadriceps and hamstring will be measured using Biodex isokinetic machine.

SECONDARY OUTCOMES:
Changes of peak VO2 | Changes of peak VO2 at 6 week
  Peak VO2 will be measured using Cosmed Quark CPET system apparatus

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No